CLINICAL TRIAL: NCT01357135
Title: Observational Study of the Treatment and Follow-up of Patients With Type II Diabetes Receiving Bitherapy With or Without Sitagliptin (Januvia®/Xelevia®).
Brief Title: An Observational Study of Type II Diabetics Treated With Dual Therapy With or Without Sitagliptin (Januvia®/Xelevia®, MK-0431-201)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0431-201
Record Dates: First submitted 2011-05-18; First posted 2011-05-20 (Estimated); Results first posted 2014-12-05 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Sitagliptin Phosphate; Sulfonylurea Compounds

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Metformin + Sitagliptin: Participants taking metformin + sitagliptin (Januvia®/Xelevia®) as prescribed in routine clinical practice.
  Interventions: Drug: Metformin; Drug: Sitagliptin
- Metformin + Sulfonylurea: Participants taking metformin + sulfonylurea as prescribed in routine clinical practice. The sulfonylurea could include: gliclazide, glibenclamide, or glimepiride.
  Interventions: Drug: Metformin; Drug: Sulfonylurea
- Sitagliptin +/- Other Antihyperglycemic Medication: Participants taking sitagliptin +/- other antihyperglycemic medication (other than metformin) as prescribed in routine clinical practice. These other antihyperglycemic medications could include: insulin, glinides, sulfonylurea, glitazone, an alpha-glucosidase inhibitor, or combinations thereof.
  Interventions: Drug: Antihyperglycemic Medication

INTERVENTIONS:
Drug: Metformin
  Groups: Metformin + Sitagliptin; Metformin + Sulfonylurea
Drug: Sitagliptin
  Groups: Metformin + Sitagliptin
Drug: Sulfonylurea
  Groups: Metformin + Sulfonylurea
Drug: Antihyperglycemic Medication
  Groups: Sitagliptin +/- Other Antihyperglycemic Medication

SUMMARY:
This is an observational study to compare the effectiveness of dual therapy of Type II diabetes mellitus with metformin + sitagliptin versus metformin + a sulfonylurea in routine clinical practice in France.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes participants
* De novo treatment (first prescription or dated within the past 8 weeks) with:
* Metformin + sitagliptin dual therapy,
* Metformin + sulfonylurea dual therapy,
* Sitagliptin as part of another treatment regimen
* Participants also eligible for treatment with sitagliptin (Januvia®/Xelevia®) or a sulfonylurea.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with type II diabetes mellitus receiving a de novo prescription (for the first time or within less than 8 weeks) for dual therapy with or without Januvia®/Xelevia® or any other treatment regimen including Januvia®/Xelevia® by general practitioners in private practice under real life conditions without any additional treatment or monitoring procedures.
Sampling Method: Non-Probability Sample
Enrollment: 3453 (Actual)
Dates: Start 2009-07-15 (Actual); Primary Completion 2013-08-31 (Actual); Study Completion 2013-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Valensi P, de Pouvourville G, Benard N, Chanut-Vogel C, Kempf C, Eymard E, Moisan C, Dallongeville J. Treatment maintenance duration of dual therapy with metformin and sitagliptin in type 2 diabetes: The ODYSSEE observational study. Diabetes Metab. 2015 Jun;41(3):231-8. doi: 10.1016/j.diabet.2015.03.007. Epub 2015 May 12. PMID 25976701
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0431-201&kw=0431-201&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an observational, non-randomized, prospective, longitudinal study of participants with Type 2 diabetes mellitus treated in routine clinical practice by 1,569 primary care practitioners in metropolitan France. Study participants were enrolled from July 29, 2009 to December 31, 2010. The end of study follow-up was August 31, 2013.
Groups:
- Sitagliptin +/- Other Antihyperglycemic Medication: Participants taking sitagliptin +/- other antihyperglycemic medications (other than metformin) as prescribed in routine clinical practice. These other antihyperglycemic medications could include: insulin, glinides, sulfonylurea, glitazone, an alpha-glucosidase inhibitor, or combinations thereof.
Period: Overall Study
Arm/Group | Metformin + Sitagliptin | Metformin + Sulfonylurea | Sitagliptin +/- Other Antihyperglycemic Medication
Started | 1874 | 733 | 846
Completed | 1276 | 510 | 583
Not Completed | 598 | 223 | 263

BASELINE CHARACTERISTICS:
Population: Baseline gender data is missing for 8 participants in the Metformin + Sitagliptin group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin + Sitagliptin | Metformin + Sulfonylurea | Sitagliptin +/- Other Antihyperglycemic Medication | Total
Number analyzed (Participants) | 1874 | 733 | 846 | 3453
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.4 (10.8) | 64.2 (11.5) | 65.5 (11.3) | 63.5 (11.2)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 758 | 311 | 372 | 1441
  Male | 1108 | 422 | 474 | 2004
  Missing | 8 | 0 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Median Duration (in Months) of Initial Dual Therapy
Description: The treatment maintenance duration corresponds to the treatment maintenance and persistence duration for dual therapy combining the same agents. Withdrawal of an agent, replacement of one agent by another or addition of a third agent is perceived as a change in treatment and, hence, the end of the treatment maintenance duration for dual therapy.
Time Frame: Up to 3 years
Population: All eligible participants receiving dual therapy with metformin + sitagliptin or metformin + sulfonylurea.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Metformin + Sitagliptin: Participants taking metformin + sitagliptin as prescribed in routine clinical practice.
Arm/Group | Metformin + Sitagliptin | Metformin + Sulfonylurea
Number analyzed (Participants) | 1874 | 733
months | 43.2 [41.4 to NA] — There were insufficient number of participants with events to estimate an upper confidence limit. | 20.2 [17.0 to 25.1]

2. Primary Outcome: Percentage of Participants With Strict Changes in Initial Dual Therapy
Description: Strict changes in dual therapy were defined as withdrawal of an agent, replacement of one agent by another, or the addition of a third agent. Changes in dose level were not considered strict changes.
Time Frame: Up to 3 years
Population: All eligible participants receiving dual therapy metformin + sitagliptin or metformin + sulfonylurea.
Measure: Number; unit: Percentage of Participants
Arm/Group | Metformin + Sitagliptin | Metformin + Sulfonylurea
Number analyzed (Participants) | 1874 | 733
Percentage of Participants | 33.1 | 46.5

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: Population of participants receiving treatment with metformin + sitagliptin or metformin + sulfonylurea or sitagliptin +/- other antihyperglycemic medication.
Arm/Group | Metformin + Sitagliptin | Metformin + Sulfonylurea | Sitagliptin +/- Other Antihyperglycemic Medication
Serious Adverse Events (participants affected / at risk) | 68/1874 | 35/733 | 66/846
Other Adverse Events (participants affected / at risk) | 0/1874 | 0/733 | 0/846
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin + Sitagliptin (N=1874) | Metformin + Sulfonylurea (N=733) | Sitagliptin +/- Other Antihyperglycemic Medication (N=846)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1) | 3 (3)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis Erosive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inflammatory bowel disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal infarction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 13 (13) | 3 (3) | 6 (6)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Heptatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral pericarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Anaesthetic complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Dural tear (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Open wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood culture positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cardiac stress test (Investigations) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 4 (4)
Diabetic foot (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (4) | 1 (1) | 2 (2)
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 2 (2)
Colon cancer Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Malignant neoplasm of ampulla of vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metatases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metatases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (2)
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Prostate cancer Stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 3 (4) | 2 (2)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Vascular dementia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 1 (1)
Completed Suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic Nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Acquired diaphragmatic eventration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Angioplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Arthrodesis (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Diverticulectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Gastrectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 2 (2) | 0 (0) | 2 (2)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Spinal laminectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Toe amputation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The adverse events in this study were not systematically collected or assessed and therefore no direct comparison can be made between adverse events in the 3 study groups/arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators cannot disclose any results without sponsor's agreement, only on request of French Health Authorities as per French law.